CLINICAL TRIAL: NCT01219205
Title: Intravitreal Bevacizumab for Macular Edema Secondary to Major and Macular Branch Retinal Vein Occlusion
Brief Title: Major and Macular Branched Retinal Venous Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Ji Won Lim, Hallym Medical center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009_128
Record Dates: First submitted 2010-10-10; First posted 2010-10-13 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Macular Edema
Keywords: macular edema secondary to retinal benous occlusion
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- major branched retinal venous occlusion (Active Comparator)
  Interventions: Procedure: intravitreal bevacizumab
- macular branched retinal venous occlusion (Active Comparator)
  Interventions: Procedure: intravitreal bevacizumab

INTERVENTIONS:
Procedure: intravitreal bevacizumab — Intravitreal injections of bevacizumab were performed under sterile conditions in the operating room. a 27-gauge needle was inserted through the corneal limbus to withdraw 0.05 ml of aqueous humor and soften the globe. Then, 1.25 mg (0.05 ㎖) of bevacizumab was injected into the vitreous in the superior temporal quadrant with a 30-gauge needle that was inserted into the eye 3.5 mm from the limbus. The postoperative medications included topical antibiotics.

SUMMARY:
Although it is important in the clinical management to classify BRVO into subtypes based on the location of the occlusion (major or macular), few studies have provided such information[8,9]. The aim of this study was to evaluate the outcome of patients with macular edema due to Branch retinal vein occlusion who were treated with intravitreal bevacizumab injection and to determine the concentrations of cytokines in the aqueous humor according to the site of the occlusion.

DETAILED DESCRIPTION:
Branch retinal vein occlusion is the second most frequent major retinal vascular disease after diabetic retinopathy. One of the main reasons for visual loss in BRVO is the development of macular edema. Treatment options for BRVO include grid laser treatment, intravitreal injection of steroids, surgical procedures, and off-label treatment with intravitreal anti-vascular endothelial growth factor (VEGF) agents. During recent years, intravitreal anti-VEGF treatment with bevacizumab has been shown to efficiently reduce macular edema and improve visual acuity in numerous case series and prospective or retrospective studies.

ELIGIBILITY:
Inclusion Criteria:

* macular edema involving the center of the fovea with a minimum central macular thickness at baseline of ≥250 μm

Exclusion Criteria:

* previous vitreoretinal surgery, intravitreal injections or laser treatment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-03; Primary Completion 2009-02 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
efficacy of intravitreal bevacizumab | baseline and 12 months after initial injection
  the number on intravitreal bevacizumab during follow-up

SECONDARY OUTCOMES:
cytokine levels in aqueous humor | before intravitreal injection
  cytokine levels in aqueous humor before bevacizumab injection

CONTACTS AND LOCATIONS:
Overall Officials: Ji Won Lim, Prof, Study Chair — Hallym Medical center
Locations (1):
- Ji Won Lim, Chuncheon, Gangwon-do, South Korea